CLINICAL TRIAL: NCT01629576
Title: Finanzielle Anreize Zur Reduktion Von Übergewicht
Brief Title: Obesity and Financial Incentives
Acronym: Obesity
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rhine-Westphalia Institute for Economic Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 010902
Record Dates: First submitted 2012-06-21; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

ARMS (3):
- control group (No Intervention)
- low reward (Experimental): economic incentive
  Interventions: Other: economic incentive
- high reward (Experimental): economic incentive
  Interventions: Other: economic incentive

INTERVENTIONS:
Other: economic incentive — economic incentive for weight loss
  Arms: low reward
Other: economic incentive — economic incentive for weight loss
  Arms: high reward

SUMMARY:
Investigate whether economic incentives help obese individuals to lose weight.

ELIGIBILITY:
Inclusion Criteria:

* BMI above 30
* age between 18 anf 75
* registered residence in the German federal state of Baden-Württemberg

Exclusion Criteria:

* considerable language barriers
* pregnancy
* psychological disorders
* eating disorders
* tumor disease within last five years
* abuse of alcohol
* abuse of drugs
* serious general diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2010-03; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
bodyweight | 22 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bad Kissingen, Baden-Würrttemberg, Germany